



## Master Statistical Analysis Plan Checklist for Investigator Initiated Trials

Phase II Trial of Eribulin in Patients Who Do Not Achieve Pathologic Complete Response (pCR) Following Neoadjuvant Chemotherapy

Sponsor: Sarah Cannon Development Innovations

(Innovations)

Study Drug: ERIBULIN

Protocol Number: BRE 186

Prepared By: Innovations



REFERENCE SOP: CDS-0102

## Statistical Analysis Plan Checklist for Investigator Initiated Trials History of Changes

This document has undergone the following changes:

| Version Number | Version Date | Description of Changes |
|----------------|--------------|------------------------|
| 1.0 | 03APR2018 | Original document |

Version 1.0, 07 JUN 2017 





REFERENCE SOP: CDS-0102

## **Statistical Analysis Plan Checklist Review and Approval**

| Approved By: | |
|-----------------------------------------|------|
| Innovations Biostatistician | Date |
| David Moorman | |
| Innovations<br>Managerial Peer-Reviewer | Date |
| Innovations Tier 1 Manager | Date |
| Innovations<br>Study Chair | Date |






| 1.1 Objectives | | |
|---|---|---|
| Primary Objective: | Assess the efficacy of eribulin when administered to patients who do not achieve pCR following standard neoadjuvant chemotherapy (+/- trastuzumab). The primary endpoint will be 2-year disease-free survival (DFS) rate. | |
| Secondary Objectives: | Assess the feasibility of administer chemotherapy and primary surgion Assess the toxicity of eribulin in the | • • |
| 1.2 Study Design | | |
| Study Type | <ul><li>☑ Non-Randomized</li><li>☐ Randomized (Allocation Ration)</li></ul> | ) |
| Details | administered postoperatively in particle and incomplete the neodiffusion of the neodif | bel trial that will evaluate 6 cycles of eribulin atients who do not achieve pCR following a standard en. There will be three cohorts of patients based on rmone-receptor-positive/HER2-negative (B), and are HER2-positive will receive trastuzumab as part of rrently with postoperative eribulin treatment. |
| | | consenting female patients who do not achieve pCR se in breast or lymph node tissue) after treatment with a apy regimen and surgery. |
| | One-hundred forty-eight patients B, and 52 in Cohort C). | will be enrolled in this trial (54 in Cohort A, 42 in Cohort |
| | All patients will receive eribulin 1.4 mg/m2 IV Days 1 and 8 every 21 days for 6 cycles. Patients with HER2-positive tumors will also receive trastuzumab 6 mg/kg IV Day 1 ever 21 days to complete a total of 1 year (52 weeks) of treatment from the start of neoadjuvant administration. If the last dose of trastuzumab was given >28 days from triatreatment start, the loading dose should be 8 mg/kg. | |
| | | n alone (Cohorts A & B) or eribulin + trastuzumab<br>status and/or hormone receptor status. |
| | Cohort | Trial Drugs & Mode of Administration |
| | Cohort A: Triple-negative | Eribulin 1.4 mg/m <sup>2</sup> IV (Days 1 & 8 every 21 days) |
| | Cohort B: Hormone-receptor-positive/HER2-negative | Eribulin 1.4 mg/m² IV (Days 1 & 8 every 21 days) |
| | Cohort C: HER2-positive | Eribulin: 1.4 mg/m² IV (Days 1 & 8 every 21 days) |
| | | Trastuzumab: 6 mg/kg IV (Day 1 every 21 days) |
| 1.3.2 Randomization | | |
| Randomization Type: | ☐ Open-Label ☐ Single B | lind Double-Blind |
| 1.4 Timing of Analysis | | |
| Planned Interim Analysis | ☐ Cohort Review / Dose Escalation | |






REFERENCE SOP: CDS-0102

| | ☐ Safety Review |
|---|---|
| | ☐ Interim Efficacy/Safety Analysis |
| | ☐ Independent DMC/DSMB |
| | ☐ Annual Report / Investigator Brochure (IB) |
| | ☐ Abstract / Scientific Presentation (Oral/Poster) |
| Final Analysis | The final analysis will occur following the completion of the trial. |
| 1.5 Responsibilities | |
| Trial Statistician: | Prepare SAP checklist and TFL shells. |
| | Review deliverables produced by statistical programmers. |
| PK Statistician: | N/A |
| Independent Statistician: | N/A |
| 1.6 Analysis Software | |
| Main statistical analysis: | SAS Version 9.3 or above |
| Other analysis software: | N/A |






| 1.7 Coding | |
|---|---|
| <ul><li>☑ Adverse Events</li><li>☐ Medical History</li></ul> | <ul> <li>MedDRA: ☐ Version</li> <li>☐ Most current release and update coding with new major releases</li> <li>☑ NCI-CTCAE Version 4.03</li> </ul> |
| <ul><li>☐ Concomitant Medication</li><li>☐ Prior Therapy</li><li>☐ Subsequent/Further Therapy</li></ul> | ☐ WHO-Drug: ☐ Version ☐ Most current release and update coding with new major releases |
| 3 Analysis Set | |
| Response Evaluable Analysis<br>Set definition: | <ul> <li>☑ All patients who have started treatment in the study</li> <li>☐ All patients who have been randomized in the study, regardless of whether they have received any treatment or not</li> <li>☐ All patients who have been randomized and have started treatment in the study</li> <li>☐ Other definition, specify:</li> </ul> |
| Per Protocol (PP) Analysis Set to be used in analysis: | ☐ Yes ☐ No If yes, please specify the criteria for exclusion from the PP population: |
| Safety (SAF) Analysis Set definition | <ul> <li>☑ All patients who have started treatment in the study. Patients will be analyzed according to the actual treatment they have received.</li> <li>☐ Other definition, specify:</li> </ul> |
| Other Analysis Set definition: | Note: Cohorts for TFLs will be: Cohort A: Triple-negative Cohort B: Hormone-receptor-positive/HER2-negative Cohort C: HER2-positive |
| 4 Baseline Value Definitions | |
| | Last value prior to first study drug treatment. |
| 5/6 Efficacy | |
| Response Criteria Used: | ☐ RECIST 1.0 ☐ RECIST 1.1 ☐ Cheson 2007 ☐ Modified RECIST – specify: ☐ Other criteria, Specify: Complete staging work-up to confirm localized disease should include computed tomography (CT) scans of the chest and abdomen/pelvis (abdomen/pelvis preferred; abdomen accepted), a CT scan of the head or MRI of the brain (if symptomatic), and either a positron emission tomography (PET) scan or a bone scan. (Note: a PET/CT is acceptable for baseline imaging in lieu of CT examinations or bone scan). Negative scans performed prior to the initiation of neoadjuvant therapy, or at any subsequent time, are acceptable and do not need to be repeated. |






Efficacy Assessment Timepoints:

REFERENCE SOP: CDS-0102

Patients will be followed every 3 months during years 1 and 2 for toxicity and disease progression.


Template ID: ASSOC-DOC-116-SOP [B]





| Efficacy Endpoints: | | | | T | |
|---|---|---|---|---|---|
| | | Endpoint | Primary Analysis<br>Population | Other Ana<br>Populatio | |
| | Primary | Disease-Free<br>Survival (DFS) | Response<br>Evaluable Analysis<br>Set | | |
| | Secondary | NA | | | |
| Definition of Terms: | | | | | |
| Response | <ul> <li>☐ Complete Response + Partial Response</li> <li>☐ Complete Response + Partial Response, confirmed with weeks apart.</li> <li>☐ Other criteria, specify:</li> </ul> | | | | |
| ☐ Clinical Benefit | Complete F | Response + Partial Respo | nse + Stable Disease | as best obs | served |
| | Complete F | Response + Partial Respo<br>ase (at least week | nse (confirmed with s from start of treatme | | s apart) + |
| | ☐ Other criteria, specify: | | | | |
| □ Progression □ | As reported by investigator | | | | |
| ☐ Subsequent Therapy | | | | | |
| ☐ Treatment Failure | | | | | |
| ☑ Duration of Follow-up | Defined as time from first treatment to death or date last known alive, reported in months | | | | |
| Definition of Endpoints: | Start Date: | Date of Randomization | □ Date of First Tr □ Date of Fir | reatment | |
| | End Date (spe | cify for all pertinent endpo | oints): | | |
| | Disease-Free Su | rvival: Event = Progression | or Death | | |
| | | Situation | Date of Event or | Censoring | Outcome |
| | No baseline as | sessment | Date of first treat | ment | Censored |
| | Progression do | ocumented | Date of progressi | on | Event |
| | Death | | Date of death | | Event |
| | No progression | n or death | Date last known a | alive | Censored |
| | Initiation of no | on-protocol anticancer there | Date of subseque therapy | ent | Censored |
| | No progression therapy | n, death, or subsequent | Date last known a | alive | Censored |




| ☐ Overall Response Rate (ORR) | Default: Estimates of rates in each treatment arm |
|---|---|
| ☐ Disease Control Rate (DCR) | ☐ Rate & 95% confidence interval (both asymptotic normal approximation and exact binomial) |
| ☐ Clinical Benefit Rate (CBR) | p-value, specify statistical test: |
| ☐ Early Progression Rate (EPR) | |
| ☐ Time To Progression (TTP) | Default: Estimates of medians (DFS) |
| ☑ Disease-Free Survival (DFS) | ☑ Other quartiles or percentages of survival required, specify: DFS estimation in 6-month increments |
| Overall Survival (OS) | ☐ Hazard ratio & 95% confidence interval between treatment arms, unstratified |
| ☐ Duration of Response | p-value, specify statistical test: |
| | Hazard ratio & 95% confidence interval between treatment arms, stratified (specify |
| ☐ Duration of Stable Disease | stratification factor(s)): |
| ☐ Time To Treatment Failure (TTF) | p-value, specify statistical test: |
| Other, Specify: | |
| 7 Safety | |
| Adverse Events | Definition of Treatment-Emergent Adverse Event (TEAE): any adverse event (AE) that starts or worsens after the start of the first dose of study treatment up to 30 days post last dose. |
| | Frequency and severity of AEs. Worst grade per patient for select AEs: related AEs by maximum grade by cohort |
| Laboratory Data | Data will be summarized by: |
| | ☐ NCI-CTCAE for CTCAE-gradable parameters, and H/L for non-CTCAE-Gradable parameter |
| | ☐ H/L for all lab parameters |
| | Worst grade per patient for select labs |

## Tier 1 Study - Tables, Figures & Listings

| Standard . | Standard TFLs | | |
|---|---|---|---|
| Table No Description | | Variables/Analyses To Be Included | Analysis Set |
| Table 1 | Disease-free Survival | Kaplan-Meier Number of patients with events, Number of patients censored, Median disease-free survival [months (95% CI)] Probability of events at: 6 month increments | Response Evaluable<br>Analysis Set |






REFERENCE SOP: CDS-0102

| Standard <sup>-</sup> | TFLs | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Analysis Set |
| Table 2 | Duration of Follow-up | Continuous numeric: N Mean Standard deviation Median Minimum Maximum | Safety Analysis Set |
| Table 3 | Treatment-related Adverse Events by Maximum Reported CTCAE Grade | by Maximum CTCAE Grade, per Cohort | Safety Analysis Set |

| Figure<br>No | Description | Variables/Analyses To Be Included | Analysis Set |
|---|---|---|---|
| Figure 1a | Disease-Free Survival – Cohort A | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | Response Evaluable<br>Analysis Set |
| Figure 1b | Disease-Free Survival – Cohort B | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | Response Evaluable<br>Analysis Set |
| Figure 1c | Disease-Free Survival – Cohort C | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | Response Evaluable<br>Analysis Set |

| | Listing<br>No. | Variables/Analyses To Be<br>Included | Analysis Set |
|---|----------------|--------------------------------------|--------------|
| ĺ | | | |
